CLINICAL TRIAL: NCT05523765
Title: A Phase 2 Randomized, Double-Masked, Dose-Ranging Study to Investigate the Safety and Efficacy of Oral Brepocitinib in Adults With Active Non-Infectious Intermediate-, Posterior-, and Panuveitis
Brief Title: A Study of Brepocitinib in Adults With Active Non-Infectious Non-Anterior Uveitis
Acronym: NEPTUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Priovant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PVT-2201-201
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Non-infectious Intermediate Uveitis; Non-infectious Posterior Uveitis; Non-infectious Pan Uveitis
Keywords: Brepocitinib; PF-06700841; uveitis; NIU
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brepocitinib Dose Level 1 by mouth (PO) once daily (QD) (Experimental)
  Interventions: Drug: Brepocitinib
- Brepocitinib Dose Level 2 by mouth (PO) once daily (QD) (Experimental)
  Interventions: Drug: Brepocitinib

INTERVENTIONS:
Drug: Brepocitinib — Oral Brepocitinib

SUMMARY:
This study will evaluate the clinical safety and efficacy of oral brepocitinib in participants with active intermediate, posterior, or pan non-infectious uveitis (NIU).

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (18-74 years old)
2. Diagnosis of non-infectious uveitis (intermediate uveitis, posterior uveitis, or panuveitis).
3. Active uveitic disease as defined by the presence of at least 1 of the following parameters in at least 1 eye, as determined by the investigator:

   1. Active, inflammatory chorioretinal and/or retinal vascular lesion; OR
   2. ≥2+ vitreous haze grade (NEI/SUN criteria).
4. Receiving up to one non-corticosteroid, non-biologic, immunomodulatory therapy
5. Weight > 40 kg with a body mass index < 40 kg/m2.

Exclusion Criteria:

1. Has isolated anterior uveitis.
2. Has confirmed or suspected current diagnosis of infectious uveitis
3. History of:

   * Any lymphoproliferative disorder
   * Active malignancy;
   * History of cancer within 5 years prior to screening (exceptions for basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of the breast, carcinoma in situ of the uterine cervix, or thyroid carcinoma.)
4. At risk of thrombosis and cardiovascular disease
5. Have a high risk for herpes zoster reactivation
6. Have active or recent infections

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Screening up to 28 days after the last dose of study drug at 52 weeks
  Safety assessments will consist of monitoring and recording all adverse events (AEs) and SAEs, laboratory evaluation for hematology, blood chemistry, and urinalysis; vital signs; electrocardiograms (ECGs); and physical examinations. The investigator will determine whether the change is clinically meaningful.

SECONDARY OUTCOMES:
Proportion of participants meeting treatment failure criteria on or after Week 6 up to Week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Johnson, PhD, Study Director — SVP, Early Development
Locations (15):
- United States (15):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Palo Alto, California
  - Clinical Trial Site, Pasadena, California
  - Clinical Trial Site, Lakewood, Colorado
  - Clinical Trial Site, Waltham, Massachusetts
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Palisades Park, New Jersey
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Eugene, Oregon
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Bellaire, Texas
  - Clinical Trial Site, Katy, Texas
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Priovant Therapeutics will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) from eligible studies upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Data requests will be reviewed and approved on the basis of scientific merit.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA). Further details on Priovant Therapeutics' data sharing criteria and process for requesting access can be obtained by emailing info@priovanttx.com.